CLINICAL TRIAL: NCT02762513
Title: Phase II Expansion Trial Evaluating Axitinib in Patients With Unresectable Recurrent, or Metastatic Head and Neck Cancer Utilizing Choi Response Criteria Phase
Brief Title: Expansion Trial for Axitinib In Head And Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2016.040; HUM00114022 (Other: University of Michigan)
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axitinib (Experimental): Participants will receive 5 mg of Axitinib twice a day continuously, with subsequent dose escalation to 7 mg and then 10 mg twice a day in the absence of grade 2 or worse toxicities
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib

SUMMARY:
This study will be a prospective, single-institution, single-arm phase II study of Axitinib in patients with unresectable recurrent and metastatic head and neck squamous cell carcinoma. The subjects will be started on treatment with 5 mg of Axitinib twice a day continuously, with subsequent dose escalation to 7 mg and then 10 mg twice a day in the absence of grade 2 or worse toxicities. This will be followed by clinical and/or radiologic response assessment after 8 weeks and subsequently every 2 months until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented squamous cell head and neck cancer with or without metastases, not amenable to curative treatment; or the patient has documented refusal of curative treatment.
* Presence of measurable disease per protocol.
* Adequate bone marrow, hepatic, and renal function.
* Age ≥18 years.
* ECOG (Eastern Cooperative Oncology Group scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 5 where 0 represents perfect health and 5 represents death.) performance status of 0-2.
* Life expectancy of ≥12 weeks.
* No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 30 minutes apart. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment.
* Signed and dated informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, including willingness to take Axitinib, laboratory tests, and other study procedures.
* If a curative treatment option in the form of chemoradiation exists in a patient with unresectable disease, this has to be attempted first and must have failed, unless the patient has documented refusal of curative treatment.

Exclusion Criteria:

* Central lung lesions involving major blood vessels (arteries or veins) or a tumor encasing major blood vessels (i.e. carotid artery).
* Active hemoptysis
* Gastrointestinal abnormalities causing impaired absorption requiring intravenous alimentation, prior surgical procedures affecting absorption including gastric resection, treatment for active peptic ulcer disease in the past 6 months, active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy, malabsorption syndromes.
* Previous treatment with anti-angiogenesis agents including thalidomide, or inhibitors of epidermal growth factor (EGF), platelet derived growth factor (PDGF), or fibroblast growth factors (FGF) receptors within 30 days preceding study entrance.
* Current use or anticipated inability to avoid use of drugs that are known potent CYP3A4/5 inhibitors
* Current use or anticipated inability to avoid use of drugs that are known CYP3A4/5 inducers
* Active seizure disorder or evidence of untreated or progressive brain metastases, spinal cord compression, or carcinomatous meningitis (Subjects with brain metastases are eligible if they have been treated and there is no CT or MRI evidence for at least 4 weeks after CNS (Central Nervous System) metastasis treatment is complete.).
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment.
* History of a malignancy (other than head and neck cancer) except those treated with curative intent for skin cancer (other than melanoma), in situ breast or in situ cervical cancer, or those treated with curative intent for any other cancer with no evidence of disease for 2 years.
* Major surgery <4 weeks or radiation therapy <2 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Patients (male and female) having procreative potential who are not willing or not able to use adequate contraception or practicing abstinence
* Women who are pregnant or breast-feeding.
* Patients with history of bleeding diathesis, arterial thromboembolism, current use of therapeutic anticoagulation with oral vitamin K antagonists, factor Xa inhibitors, heparin products, oral direct thrombin inhibitors, or presence of non-healing wounds. Low-dose anticoagulants for maintenance of patency of central venous access device or prevention of deep venous thrombosis is allowed.
* Patients residing in prison.
* Prior experimental therapy within 30 days of planned start of this trial.
* HIV virus infection irrespective of viral load, treatment status, or CD4 count, or acquired immunodeficiency syndrome (AIDS)-related illness. HIV testing is not required by this protocol.
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
* History of deep vein thrombosis or pulmonary embolism within 6 month of anticipated starting of Axitinib.
* Availability of curative treatment option for the patient's cancer, whether surgery, chemotherapy, radiation, or combination thereof, unless the patient has documented refusal of curative treatment.
* Increased risk of wound dehiscence or presence of non-healing wounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Swiecicki, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient enrolled but progressed before starting study treatment.
Period: Overall Study
Arm/Group | Axitinib
Started (Started study treatment with axitinib) | 28
Completed (Completed at least one 28-day cycle of treatment with axitinib.) | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 28
Age, Continuous [Mean (Full Range); unit: years] | 63.9 [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28
ECOG performance status [Count of Participants; unit: Participants]
  0 (fully functional) | 11
  1 (minor impairment) | 17
Disease primary site [Count of Participants; unit: Participants]
  Oral cavity | 2
  Oropharynx | 13
  Larynx | 4
  Nasopharynx | 3
  Cutaneous | 6
HPV status [Count of Participants; unit: Participants]
  Positive | 10
  Negative | 17
  Unknown | 1
Previous lines of therapy [Count of Participants; unit: Participants]
  0 | 11
  1 | 6
  2 | 5
  >=3 | 6
Previous exposure to platinum [Count of Participants; unit: Participants]
  Sensitive | 11
  Refractory | 17
Previous exposure to PD-1 inhibitor [Count of Participants; unit: Participants] — Population: Only patients with previous exposure to PD-1 inhibitor are included in this measure (n=11)
  Participants
    number analyzed (Participants) | 11
    Primary resistant | 3
    Acquired resistance | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Evaluable Patients Alive at 6 Months
Description: Evaluable defined as any participant who receives at least one cycle of Axitinib. Number of evaluable patients and percentage of patients alive at 6 months is reported.
Time Frame: 6 Months after treatment initiation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 28
percentage of participants | 71 [53 to 85]

2. Secondary Outcome: Median Overall Survival Time
Description: median will be calculated by Kaplan-Meier method.
Time Frame: Up to approximately 2.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib
Number analyzed (Participants) | 28
months | 9.8 [5.9 to 12.2]
Statistical Analysis 1: Comparison: Axitinib; Test type: Other; Median overall survival time (months) = 9.8 — Median calculated by Kaplan-Meier method

3. Secondary Outcome: Median Progression Free Survival (PFS) Time
Description: Median will be calculated by Kaplan-Meier method.
Time Frame: Up to approximately 2.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib
Number analyzed (Participants) | 28
months | 3.5 [2.4 to 5.4]
Statistical Analysis 1: Comparison: Axitinib; Test type: Other; Median PFS time (months) = 3.5 — Median calculated by Kaplan-Meier method

4. Secondary Outcome: Best Overall Response
Description: Tabulation of best response measured by Choi. Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progression (PD) at 16 weeks. CR is defined as no new lesions and the disappearance of all lesions. PR is defined as a decrease in size of ≥ 10% or a decrease in tumor density (HU) ≥ 15% on CT (Computerized Tomography), no new lesions and no obvious progression of non-measurable disease
Time Frame: 16 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 28
Participants
  Progressive disease | 10
  Stable disease | 3
  Partial response | 11
  Complete response | 1
  Off treatment before 8-wk scan | 3

5. Secondary Outcome: The Number of Patients That Experience Grade 3 or Worse Toxicities
Description: Assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. For any treatment-related toxicity that occurred at any grade with a frequency greater than 10% in the overall study population, grade 3 or worse toxicities are shown here.
Time Frame: Duration of treatment and up to 28 days after treatment discontinuation
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 28
Participants
  Fatigue | 6
  Hypertension | 2
  Oral mucositis | 2
  Diarrhea | 1
  Oral pain | 1
  Bleeding | 1

ADVERSE EVENTS:
Time Frame: AEs were collected from time of initial study treatment administration through death or 28 days after treatment discontinuation. Median treatment duration was three 28-day cycles (range 1-9 cycles). All-cause mortality data was collected from time of initial study treatment administration through death or up to 36 months after treatment discontinuation. Median follow-up was 18 months (range 1-36).
Arm/Group | Axitinib
All-Cause Mortality (participants affected / at risk) | 20/28
Serious Adverse Events (participants affected / at risk) | 8/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib (N=28)
Cardiac arrest (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib (N=28)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (4)
Eye disorders - Other (Eye disorders) | 2 (2)
Eye pain (Eye disorders) | 1 (1)
Papilledema (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 8 (10)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 4 (9)
Nausea (Gastrointestinal disorders) | 10 (10)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 4 (4)
Rectal perforation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Edema face (General disorders) | 1 (1)
Fatigue (General disorders) | 21 (46)
Neck edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3)
Pain (General disorders) | 7 (7)
Papulopustular rash (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Blood bilirubin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 7 (9)
Anorexia (Metabolism and nutrition disorders) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (2)
Brachial plexopathy (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 5 (6)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertension (Vascular disorders) | 15 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT02762513/Prot_SAP_000.pdf